CLINICAL TRIAL: NCT04453150
Title: Ketone Bodies and Gut Microbiota Role in the Dietetic Approach of Obesity
Brief Title: Microbiota in Dietary Approach to Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISCIII CP18/01160
Record Dates: First submitted 2020-04-17; First posted 2020-07-01 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2021-07

CONDITIONS: Obesity
Keywords: Ketosis; Microbiota
MeSH Terms: conditions — Obesity; Ketosis | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Standard hypocaloric diet (Experimental): Mediterranean diet based on olive oil as main fat and regular consumption of vegetables (2 daily rations), fruits 3 daily rations), legumes (3 weekly rations), fish (3 weekly rations), with low consumption of red meat and meat products (less than twice a week), dairy foods (less than once a week) and no sweets, pastries or sugary drinks. Diet will produce a 600 kcal per day caloric deficit, according to the Harris-Benedict equation for each subject. Diet will include 45% carbohydrates, 35% fat, 20% protein distributed in at least 4 meals (breakfast, lunch, afternoon snack and dinner).
  Interventions: Other: Standard hypocaloric die
- Intermittent fasting 16/8 (early fasting) (Experimental): Diet will produce a 600 kcal per day caloric deficit, according to the Harris-Benedict equation for each subject. Diet will include 45% carbohydrates, 35% fat, 20% protein, but it will be consumed for 8 hours a day (from 12 am. to 8 pm.), maintaining 16 fasting hours (from 8 pm. to 12 am. the following day).
  Interventions: Other: Intermittent fasting 16/8 (early fasting)
- Intermittent fasting 16/8 (late fasting) (Experimental): Diet will produce a 600 kcal per day caloric deficit, according to the Harris-Benedict equation for each subject. Diet will include 45% carbohydrates, 35% fat, 20% protein, but it will be consumed for 8 hours a day (from 8 am. to 4 pm.), maintaining 16 fasting hours (from 4 pm. to 8 am. the following day).
  Interventions: Other: Intermittent fasting 16/8 (late fasting)
- Alternate-day fasting (Experimental): In this diet subjects alternate norm caloric diet during 24 h (according to Harris-Benedict equation) and a diet including only 25% of caloric requirements the following 24 h (this day diet will include 5 % carbohydrates, 65% fat and 30% high biological value protein).
  Interventions: Other: Alternate-day fasting
- Ketogenic diet (Experimental): Diet will produce a 600 kcal per day caloric deficit, according to the Harris-Benedict equation for each subject. Diet will include 5 % carbohydrates, 65% fat and 30% high biological value protein.
  Interventions: Other: Ketogenic diet

INTERVENTIONS:
Other: Standard hypocaloric die — Standard hypocaloric diet
  Arms: Standard hypocaloric diet
Other: Intermittent fasting 16/8 (early fasting) — Intermittent fasting 16/8 (early fasting)
  Arms: Intermittent fasting 16/8 (early fasting)
Other: Intermittent fasting 16/8 (late fasting) — Intermittent fasting 16/8 (late fasting)
  Arms: Intermittent fasting 16/8 (late fasting)
Other: Alternate-day fasting — Alternate-day fasting
  Arms: Alternate-day fasting
Other: Ketogenic diet — Ketogenic diet
  Arms: Ketogenic diet

SUMMARY:
Main aim: Study the anthropometric, metabolic, cardiovascular and neurocognitive and gut microbiota changes of different approaches for the weight reduction that increase the ketone bodies in a different proportion in relation to the classic hypocaloric diet.

Objective 1: Study the effect of hypocaloric diets that increase the ketone bodies on gut microbiota and its relationship with anthropometric changes and of the Brown adipose tissue, Objective 2: with the metabolic and inflammatory changes, Objective 3: on the cardiovascular system, Objective 4: on the neurocognition, Objective 5: if they are associated to epigenetic changes that may explain the changes found in the other objectives. Objective 6: Determine the safety of the diets that increase the ketone bodies compared to the classic hypocaloric diet, Objective 7: if the effects of the different dietary approaches are maintained during the medium time, and Objective 8: Verify in experimental models (microbiota transplants from humans with different diets to germ-free mice, ketosis dietary models, and ketone bodies administration) the causality of the gut microbiota of these findings.

Methodology: Model 1: Dietary intervention in humans with 4 types of diet with a different increase of the ketone bodies: classic hypocaloric diet (DH); diet with 8h of feeding and 16h of starving in periods of 24h (D16); diet with intermittent caloric restriction (DA); and normal in protein and low in carbohydrates hypocaloric ketogenic diet (DC).

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI≥30-45 kg/m2)

Exclusion Criteria:

* Type 2 diabetes mellitus
* Patients with major cardiovascular events in the 6 months prior to the study beginning.
* Previous or current history of inflammatory disease.
* Active infectious disease.
* The refusal of the patient to participate in the study
* Consumption of probiotics or prebiotics
* Antibiotic therapy in the 3 months prior to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota composition | Baseline, 12 weeks
  To evaluate changes in gut microbiota composition from baseline using different strategies for weight loss which increase ketone bodies in comparison to a standard hypocaloric diet. Change from baseline in 16S rRNA amplicons of fecal community DNA at 3 months and 6 months

SECONDARY OUTCOMES:
Changes in weight | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies on anthropometric parameters in comparison to a standard hypocaloric diet
Changes in body mass index. | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies on body mass index in comparison to a standard hypocaloric diet
Changes in waist circumference. | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies on the waist circumference in comparison to a standard hypocaloric diet
Changes in body composition. | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies on anthropometric parameters in comparison to a standard hypocaloric diet measured by bioelectrical impedance analysis
Changes in brown adipose tissue. | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies on brown adipose tissue in comparison to a standard hypocaloric diet, measured by Positron emission tomography with 18F-fluorodeoxyglucose (18F-FDG PET).
Changes in uncoupling protein 1 (UCP1) | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies on brown adipose tissue UCP1 in comparison to a standard hypocaloric diet using a sample of subcutaneous white adipose tissue assessed by mRNA qPCR.
Changes in physical activity. | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies on physical activity in comparison to a standard hypocaloric diet measured by accelerometry
Changes in blood pressure | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies over the cardiovascular system in comparison to a standard hypocaloric diet based on blood pressure
Changes in the punctuation in neurocognitive test | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies on neurocognition, in comparison to a standard hypocaloric diet, measured by neurocognitive test
Changes in heart rate | Baseline, 12 weeks
  To analyze the effect of hypocaloric diets which increase ketone bodies on heart function measured by heart rate in comparison to a standard hypocaloric diet, measured by Holter.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J. Tinahones, PhD, Principal Investigator — Instituto de Investigacion Biomedica de Malaga
Locations (1):
- Virgen de la Victoria Hospital, Málaga, Spain

REFERENCES:
- [Derived] Martinez-Montoro JI, Bandera B, Gutierrez-Bedmar M, Gomez-Perez AM, Macias-Gonzalez M, Moreno-Indias I, Tinahones FJ. Effect of a ketogenic diet, time-restricted eating, or alternate-day fasting on weight loss in adults with obesity: a randomized clinical trial. BMC Med. 2025 Jul 1;23(1):368. doi: 10.1186/s12916-025-04182-z. PMID 40598397
- [Derived] Mela V, Heras V, Iesmantaite M, Garcia-Martin ML, Bernal M, Posligua-Garcia JD, Subiri-Verdugo A, Martinez-Montoro JI, Gomez-Perez AM, Bandera B, Moreno-Indias I, Tinahones FJ. Microbiota fasting-related changes ameliorate cognitive decline in obesity and boost ex vivo microglial function through the gut-brain axis. Gut. 2025 Oct 8;74(11):1828-1846. doi: 10.1136/gutjnl-2025-335353. PMID 40335161